CLINICAL TRIAL: NCT02757729
Title: Multi Center, Randomized, Double-blind, Placebo-controlled Parallel-group, Phase II Clinical Trial to Evaluate the Safety and Efficacy of PAC-14028 Cream in Mild to Moderate Atopic Dermatitis Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-TRPV1-PII_04
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PAC-14028 cream 0.1% (Experimental): PAC-14028 cream 0.1%, Twice daily for 8 weeks
  Interventions: Drug: PAC-14028 cream 0.1%
- PAC-14028 cream 0.3% (Experimental): PAC-14028 cream 0.3%, Twice daily for 8 weeks
  Interventions: Drug: PAC-14028 cream 0.3%
- PAC-14028 cream 1.0% (Experimental): PAC-14028 cream 1.0%, Twice daily for 8 weeks
  Interventions: Drug: PAC-14028 cream 1.0%
- PAC-14028 cream vehicle (Placebo Comparator): PAC-14028 cream vehicle, Twice daily for 8 weeks
  Interventions: Drug: PAC-14028 cream vehicle

INTERVENTIONS:
Drug: PAC-14028 cream 0.1% — Topical application
  Arms: PAC-14028 cream 0.1%
Drug: PAC-14028 cream 0.3% — Topical application
  Arms: PAC-14028 cream 0.3%
Drug: PAC-14028 cream 1.0% — Topical application
  Arms: PAC-14028 cream 1.0%
Drug: PAC-14028 cream vehicle — Topical application
  Arms: PAC-14028 cream vehicle

SUMMARY:
This is a phase 2 study to investigate the safety and efficacy of PAC-14028 cream in Atopic Dermatitis patients.

DETAILED DESCRIPTION:
PAC-14028 Cream (0.1%, 0.3%, 1.0%) or placebo will be treated to Mild to Moderate Atopic Dermatitis patients twice daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 19 - 70 years.
* Who was diagnosed with Atopic Dermatitis according to Haniffin and Rajka criteria.
* Whose affected BSA is over 5% and IGA score is 2 (mild) to 3 (moderate).
* Who voluntarily agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

* Who has skin diseases other than atopic dermatitis or scar in the affected area which can affect the study, determined by the study investigators.
* Who has clinically significant medical history or diseases involving liver, kidney, neurological system, psychical disorder that can affect study results.
* Who has used systemic steroids, antibiotics, immunosuppressants, or received photochemical therapy within 28 days before study drug administration.
* Who has used topical steroids, immunosuppressants or antibiotics to treat atopic dermatitis within 14 days before study drug administration.
* Who has used or is expected to inevitably use prohibited concomitant medications during the study.
* Women who is pregnant /breast-feeding, or who has childbearing potential and does not use available contraceptives.
* Who has dosed other study medications within 30 days before screening.
* Who is determined ineligible for study participation by investigators for any other reasons.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Success rate of Investigator's Global Assessment (IGA) | 8 weeks
  percent of patients with IGA score of 0 (clear) or 1 (almost clear)

SECONDARY OUTCOMES:
Success rate of Investigator's Global Assessment (IGA) | 1, 3, 6 week(s)
  percent of patients with IGA score of 0 (clear) or 1 (almost clear)
Change in SCORAD (Severity Score of Atopic Dermatitis) | 1, 3, 6, 8 week(s)
% Change in Eczema Area and Severity Index (EASI) | 1, 3, 6, 8 week(s)
Success rate of Pruritus Severity score | 1, 3, 6, 8 week(s)

CONTACTS AND LOCATIONS:
Overall Officials: Beomjoon Kim, MD, PhD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No